CLINICAL TRIAL: NCT00709527
Title: A Phase 1 Ascending Dose And Parallel Group Trial To Establish The Safety, Tolerability And Pharmacokinetic Profile of Multiple Intravitreous Injections of ARC1905 (Anti-C5 Aptamer) Given In Combination With Multiple Doses of Lucentis® 0.5 mg/Eye In Subjects With Neovascular Age-Related Macular Degeneration
Brief Title: ARC1905 (Anti-C5 Aptamer) Given With Lucentis 0.5 mg In People With Neovascular Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ophthotech Corporation (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPH2000
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: AMD

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Avacincaptad Pegol

INTERVENTIONS:
Drug: Avacincaptad Pegol — intravitreal injection
  Other Names: Zimura (previous name); IZERVAY; ARC1905

SUMMARY:
The objectives of this study are to evaluate the safety, tolerability, and pharmacokinetic profile of multiple doses of ARC1905 intravitreous injection when administered in combination with multiple doses of Lucentis® 0.5 mg/eye, or with one induction dose of Lucentis 0.5 mg/eye in subjects with subfoveal choroidal neovascularization secondary to age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Subfoveal choroidal neovascularization (CNV) due to AMD (i.e., predominately classic, minimally classic or occult no classic) as documented by fluorescein angiogram.

Exclusion Criteria:

* Previous or concomitant therapy with intravitreous corticosteroids.
* Any of the following underlying diseases including:
* Diabetic retinopathy
* History or evidence of severe cardiac disease (e.g., NYHA Functional Class III or IV), history or clinical evidence of unstable angina, acute coronary syndrome, myocardial infarction or revascularization within last 6 months, ventricular tachyarrythmias requiring ongoing treatment.
* History or evidence of clinically significant peripheral vascular disease, such as intermittent claudication or prior amputation.
* Clinically significant impaired renal (serum creatinine >2.5 mg/dl or s/p renal transplant or receiving dialysis) or hepatic function. Patients with results outside these ranges may be enrolled in consultation with Ophthotech.
* Stroke (within 12 months of trial entry).
* Any major surgical procedure within one month of trial entry.
* Previous therapeutic radiation in the region of the study eye.
* Any treatment with an investigational agent in the past 60 days for any condition.
* Women who are pregnant or nursing.
* Known serious allergies to the fluorescein dye used in angiography, to the components of the ranibizumab formulation, or to the components of the ARC1905 formulation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-10-16 (Actual); Primary Completion 2009-12-30 (Actual); Study Completion 2009-12-30 (Actual)

PRIMARY OUTCOMES:
Presence of any dose-limiting toxicity (DLT), safety endpoints include adverse events, vital signs, ophthalmic variables and outcomes | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthotech Corp, New York, New York, United States

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=26387&tenant=MT_AST_9011